CLINICAL TRIAL: NCT04993248
Title: Nursing Intervention "Dialogue Circles" to Reduce the Level of Caregiver Overload in Complex Chronic Patients and Advanced Chronic Disease
Brief Title: "Dialogue Circles" to Reduce the Level of Caregiver Overload in Complex Chronic Patients and Advanced Chronic Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20/112-PCV
Record Dates: First submitted 2021-07-13; First posted 2021-08-06 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-07

CONDITIONS: Caregiver Burnout
Keywords: Informal caregiver; Overload; Nurse
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Masking Description: Single masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will offer participants the opportunity to share feelings and needs with people who are in a similar situation to their own.
  Each intervention consists of 3 dialogue circles per group. Each group is composed of 10 participants and a facilitator, in all interventions the facilitator will be the principal investigator.
  Interventions: Other: Dialog Circle
- Control (No Intervention): Usual intervention

INTERVENTIONS:
Other: Dialog Circle — The intervention will offer participants the opportunity to share feelings and needs with people who are in a similar situation to their own.
  Each intervention consists of 3 dialogue circles per group. Each group is composed of 10 participants and a facilitator, in all interventions the facilitator will be the principal investigator.
  Arms: Intervention

SUMMARY:
The increase in life expectancy and the decrease in the birth rate have led to an aging population and a higher prevalence of chronic diseases. This has generated the need for informal caregivers of older adults to face health care situations of this population. On the other hand, it has become evident how the epidemiological profile has changed over the last 50 years, with a decrease in infectious diseases and a higher prevalence of chronic non-communicable diseases, which increase the demand for family caregivers. Caring for a dependent family member can negatively affect the caregiver's health in his or her affective and working life. In the first phase, a cross-sectional descriptive study will be carried out and in the second phase, an experimental study, randomized clinical trial (RCT) with simple masking will be conducted Objectives: Phase I general objective is to describe the sociodemographic characteristics of the study sample. Specific in this phase are to analyze the relationship between level of caregiver strain and sociodemographic variables collected from primary caregivers, to analyze the relationship between level of caregiver strain and the patient's ability to perform activities of daily living, to analyze the relationship between level of caregiver strain and the patient's ability to perform activities of daily living. To analyze the relationship between level of caregiver overload and deterioration in the patient's cognitive sphere. To analyze the relationship between overload and the instrumental activities that the patient can perform. To analyze the relationship between overload and mental health from a positive perspective. Phase II: the general objective is to determine the efficacy of the nursing intervention, dialogue circles, to reduce the level of overload perceived by caregivers of patients identified as complex chronic patients and chronic advanced disease. The specific objectives are to compare the level of overload perceived by the main caregivers before and after the intervention between the experimental group and the control group, and the degree of satisfaction with the dialogue circles nursing intervention. It will be carried out in Catalonia, in the populations of the metropolitan area of Barcelona, belonging to the Primary Care Service (SAP) Baix Llobregat Centre.

ELIGIBILITY:
Inclusion Criteria:

* - Primary caregivers of patients identified as Patient Chronic and/or advanced chronic disease who are in the case management service portfolio in the basic areas of SAP Baix Llobregat Centre and Delta de Llobregat.
* Primary caregivers with the abbreviated caregiver burden scale administered.

Exclusion Criteria:

* Caregivers under 18 years of age.
* Occasional caregivers.
* Professional or contracted caregivers.
* Primary caregivers of patients diagnosed with any type of dementia.
* Primary caregivers participating at the time of the intervention in some type of individual or group psychological intervention.
* Not wishing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Overload caregivers | Changes in the level of overload (Pre intervention and 15 days after nursing intervention )
  Short Interview on burden of care for caregivers in primary care

CONTACTS AND LOCATIONS:
Overall Officials: Jose Manuel Camarena, Principal Investigator — Idiap
Locations (1):
- Jose Manuel Tinoco Camarena, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carreño SP, Sánchez-Herrera B, Carrillo GM, Chaparro-Díaz L, Gómez OJ. Carga de la enfermedad crónica para los sujetos implicados en el cuidado. Rev. Fac. Nac. Salud Pública 2016; 34(3): 342-349.
- [Background] Martín M, Salvadó I, Nadal S, Miji LC, Rico JM, Lanz P. Adaptación para nuestro medio de la escala de sobrecarga del cuidador (Caregiver Burden Interview) de Zarit. Rev Gerontol. 1996; 6:338-46.
- [Background] 3. Sánchez Martínez RT, Molina Cardona EM,Gómez-Ortega OR. Intervenciones de enfermería para disminuir la sobrecarga en cuidadores: un estudio piloto. Revista Cuidarte. 2016; 7(1):1171-84.
- [Background] Herbert R, Bravo G, Preville M. Reliability, validity and reference values of the Zarit Burden Interview for assessing informal caregivers of community-dwelling older persons with dementia. Can J Aging 2000;19:494-507. http://dx.doi.org/10.1017/S0714980800012484
- [Background] Taub A, Andreoli SB, Bertolucci PH. Dementia caregiver burden: reliability of the Brazilian version of the Zarit caregiver burden interview. Cad Saude Publica. 2004 Mar-Apr;20(2):372-6. doi: 10.1590/s0102-311x2004000200004. Epub 2004 Apr 6. PMID 15073616
- [Result] Ankri J, Andrieu S, Beaufils B, Grand A, Henrard JC. Beyond the global score of the Zarit Burden Interview: useful dimensions for clinicians. Int J Geriatr Psychiatry. 2005 Mar;20(3):254-60. doi: 10.1002/gps.1275. PMID 15717336
- [Result] Velez Lopera JM, Berbesi Fernandez D, Cardona Arango D, Segura Cardona A, Ordonez Molina J. [Validation of the abbreviated Zarit scales for measuring burden syndrome in the primary caregiver of an elderly patient]. Aten Primaria. 2012 Jul;44(7):411-6. doi: 10.1016/j.aprim.2011.09.007. Epub 2011 Nov 4. Spanish. PMID 22055916
- [Result] Arai Y, Kudo K, Hosokawa T, Washio M, Miura H, Hisamichi S. Reliability and validity of the Japanese version of the Zarit Caregiver Burden interview. Psychiatry Clin Neurosci. 1997 Oct;51(5):281-7. doi: 10.1111/j.1440-1819.1997.tb03199.x. PMID 9413874